CLINICAL TRIAL: NCT02323152
Title: PREVENTION OF POSTPARTUM DEPRESSION DEVELOPMENT IN WOMEN WITH VERY HIGH RISK
Acronym: PROGEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, MARIA PURIFICACIÓN LOPEZ PEÑA, Maria Purificación Lopez Peña, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROGEA
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Postpartum Depression
Keywords: women; high risk
MeSH Terms: conditions — Depression, Postpartum | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- psychoeducation (Experimental): Usual treatment + psychoteraphy focused on problem solving (6 sessions). The psychoeducational programme consists of 6 sessions of 60 minutes, one per week.
  Interventions: Behavioral: psychoeducation
- Control group (Active Comparator): Puerperal control with their doctor. This group will also be interviewed with the same frecuency of the experimental group but will not receive a psichologycal treatment.
  Interventions: Other: Standard care

INTERVENTIONS:
Behavioral: psychoeducation — Usual treatment + psychoteraphy focused on problem solving (6 sessions). The psychoeducational programme consists of 6 sessions of 60 minutes, one per week.
  Arms: psychoeducation
Other: Standard care — Puerperal control with their doctor. This group will also be interviewed with the same frecuency of the experimental group but will not receive a psichologycal treatment
  Arms: Control group

SUMMARY:
Postpartum depression is a disease with a prevalence of 10% which has not only deleterious consequences for the mother but also for the baby and can delay the physical, social and cognitive development of the baby. Therefore we consider very important to prevent this disease as from the centers of care for women with a multidisciplinary approach. The aim of this study is to determine whether psychoeducation oriented in problem solving is effective in preventing the development of postpartum depression in women with very high risk.

Methodology: screening of 1000 women in 3rd trimester of pregnancy. We expect that 25% have at least one risk factor for postpartum depression (250). Of these women, aproximately a 50% will have a very high risk of developing postpartum depressión and will be included in the study (n = 125). These women will be randomized to two groups: treatment with psychotherapy focused on problem solving (6 sessions: 1 individual session + 5 group sessions) or usual care control group (usual postpartum control).

After treatment, women will be evaluated twice, at the end of therapy and at 6 weeks. Survival curves will be used tu assess the time it takes patients to develop major depression in the postpartum.

ELIGIBILITY:
Inclusion criteria

1. General criteria for inclusion in the study:

   1. Pregnant women in the 3rd quarter. In the case of inclusion of children in the study were notified each case their participation to the Department.
   2. Signature of informed consent.
2. Inclusion criteria for treatment group:

   1. Submitted one or more risk factor for developing postpartum depression:

      * Depressive or anxious pathology during pregnancy.
      * Personal history of severe mental disorder (schizophrenia and other psychoses, bipolar disorder, depressive disorder).
      * Family history of severe mental disorder.
      * Concomitant medical diseases associated with depression (diabetes, heart disease, hypertension, obesity).
      * Low or very low socioeconomic status.
      * Lack of support for women (couples, family, friends or others).
   2. Submit a score ≥7.5 in the EPDS questionnaire. According Vega-Dienstmainer (Vega-Diesnstmainer JM, 2002), there weren't women with lower score than 7.5 that had been diagnosed with DPP (sensitivity and positive predictive value of 100%). Therefore, we considered selecting those patients with higher score of 7.5 on the EPDS scale.

Exclusion criteria

1. Mental Retardation.
2. Severe mental disorder decompensation that prevents understanding of the objectives of the study.
3. Submit language difficulties that impede verbal comprehension / reading-writing.
4. Submit a major depressive episode according to DSM-IV TR (depressive symptoms of sufficient intensity and longer duration than 2 weeks).

All participants will be informed that they will be randomized to on of the two study groups and will only be included if they give their informed consent to participate in the study. Women in both groups will be evaluated at baseline (pre-intervention) at 6 and 12 weeks (postinternveción).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2012-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Depression Scale | 6 weeks
  Participants' symptoms are assessed using the Edimburg scale (Cox et al., 1987) This 10 item self report measure is designed to screen women for symptoms of emotional distress during pregnancy and the postnatal period.This scale has been validated in Castilian Spanish 2012 (CARPETA)

SECONDARY OUTCOMES:
Depression Scale | 12 weeks
  Participants' symptoms are assessed using the Edimburg scale (Cox et al., 1987) This 10 item self report measure is designed to screen women for symptoms of emotional
Vulnerable personality | 6 weeks
  The Vulnerable Personality Style Questionnaire (VPSQ) is a nine-item self-report scale developed to asses personality traits which increase the risk of postpartum depression(Gelabert et al., 2011).
Vulnerable personality | 12 weeks
  The Vulnerable Personality Style Questionnaire (VPSQ) is a nine-item self-report scale developed to asses personality traits which increase the risk of postpartum depression(Gelabert et al., 2011).
Physical Activity Questionare | 6 weeks
  IPAQ: The International Physical Activity Questionnaires (IPAQ) provides a set of well-developed instruments that can be used internationally to obtain comparable estimates of physical activity. The long version we use provide more detailed information often required in research work or for evaluation purposes (Martinez-Gonzalez et al., 2005)
  GPAC : The Global Physical Activity Questionnaire was developed by WHO for monitoring physical activity in countries. Collects information about participation in physical activity and sedentary behavior in three frames (or fields). These fields are:
  * activity at work
  * activity at displacement
  * leisure activity
Physical Activity Questionare | 12 weeks
  IPAQ: The International Physical Activity Questionnaires (IPAQ) provides a set of well-developed instruments that can be used internationally to obtain comparable estimates of physical activity. The long version we use provide more detailed information often required in research work or for evaluation purposes (Martinez-Gonzalez et al., 2005)
  GPAC : The Global Physical Activity Questionnaire was developed by WHO for monitoring physical activity in countries. Collects information about participation in physical activity and sedentary behavior in three frames (or fields). These fields are:
  * activity at work
  * activity at displacement
  * leisure activity
Temperament Style | 6 weeks
  Merrill-Palmer-Revised Scales of Development: We measure the babys temperament with the Merrill-Palmer-Revised Scales of Development. This escale evaluates five main areas of development: cognition, language, motor skills, adaptive behavior and self-care and socioemotional. Provides information on global development the child to assess the presence of possible delays in some areas (Roid et al., 2004).
Temperament Style | 12 weeks
  Merrill-Palmer-Revised Scales of Development: We measure the babys temperament with the Merrill-Palmer-Revised Scales of Development. This escale evaluates five main areas of development: cognition, language, motor skills, adaptive behavior and self-care and socioemotional. Provides information on global development the child to assess the presence of possible delays in some areas (Roid et al., 2004).

CONTACTS AND LOCATIONS:
Overall Officials: AMAIA.UGARTEUGARTE@osakidetza.net UGARTE UGARTE, Principal Investigator — Hospital Universitario Araba

REFERENCES:
- [Derived] Ugarte AU, Lopez-Pena P, Vangeneberg CS, Royo JG, Ugarte MA, Compains MT, Medrano MP, Toyos NM, Lamo EA, Duenas MB, Gonzalez-Pinto A. Psychoeducational preventive treatment for women at risk of postpartum depression: study protocol for a randomized controlled trial, PROGEA. BMC Psychiatry. 2017 Jan 13;17(1):13. doi: 10.1186/s12888-016-1162-5. PMID 28086766